CLINICAL TRIAL: NCT02990585
Title: The Effect of an 8-session Back School Versus a Single, Abbreviated Session When Looking at Non-specific Low Back Pain in an Urban Setting
Brief Title: Back School for Non-specific Low Back Pain (LBP) in an Urban Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Marie-Eve Pepin, Assistant Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 041016MP4E
Record Dates: First submitted 2016-11-09; First posted 2016-12-13 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- One individual back school session (Active Comparator): The 1 individual session will consist of a 60 min 1-on-1 education/exercise session with an athletic trainer. Information will be an abbreviated version of the 8-session school and fill focus on the strengthening, stretching, pain control and movement re-education most needed for the individual.
  Interventions: Other: Back school
- 8 group session of back school (Active Comparator): All sessions last 45-60 minutes. There will be up to 8 participants in each session which will be led by an athletic trainer or rehabilitation trainer. Pain management, prevention strategies, and active treatment will be covered in the 8 sessions. Active treatment includes strengthening, stretching, pain control, movement re-education, and walking.
  Interventions: Other: Back school

INTERVENTIONS:
Other: Back school

SUMMARY:
This study will be a comparative design between 2 groups of subjects attending classes on back education in an urban setting. Participants will be randomized to either an individual one-on-one back school session or to the 8 group sessions.

ELIGIBILITY:
Inclusion Criteria:

* Participants 18 years of age or older who have been suffering from non-specific LBP for at least 3 months

Exclusion Criteria:

* Additional impairments contraindicating their safe participation in the back school program, such as evidence of spinal cord pathology, cauda equina, progressive neurological damage, infection, inflammation, malignancy, fracture or a progressive, neurodegenerative disease as well as back surgery within the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-10; Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Change in the Modified Oswestry Disability Index | At 4 weeks, 10 weeks, 4 months, and 7 months

SECONDARY OUTCOMES:
Change in the Fear Avoidance Belief Questionnaire -Physical Activity portion | At 4 weeks, 10 weeks, 4 months, and 7 months
Change in the Numeric pain rating scale | At 4 weeks, 10 weeks, 4 months, and 7 months
Change in the International Physical Activity Questionnaire | At 4 weeks, 10 weeks, 4 months, and 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie Pepin, DPT, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No